CLINICAL TRIAL: NCT03475875
Title: Contact Lenses With New UV-blocker Manufactured With Different Techniques
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6140
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Correction of Refraction Error; Attenuation of Bright Light

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL/CONTROL (Experimental): Subjects that are of 18 years or older and current spherical soft contact lens wearers will wear the Test and Control lenses for two weeks each in random order with one of the study lenses being worn twice for a total of 6 weeks per subject.
  Interventions: Device: senofilcon A TEST Lens; Device: senofilcon A CONTROL Lens
- CONTROL/TEST/TEST (Experimental): Subjects that are of 18 years or older and current spherical soft contact lens wearers will wear the Test and Control lenses for two weeks each in random order with one of the study lenses being worn twice for a total of 6 weeks per subject.
  Interventions: Device: senofilcon A TEST Lens; Device: senofilcon A CONTROL Lens

INTERVENTIONS:
Device: senofilcon A TEST Lens — senofilcon A with new UV blocker investigational process
Device: senofilcon A CONTROL Lens — senofilcon A with new UV blocker standard process

SUMMARY:
This study is a randomized, 4-visit, double-masked, 2x3 bilateral crossover, dispensing trial. The study lenses will be worn as daily wear (DW) for a period of two weeks each with one of the study lenses being worn twice. Each study lens is expected to be worn at least five (5) days per week for at least six (6) hours per day worn. There will be no washout period between study lenses.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Healthy adult males or females age ≥18 years of age with signed informed consent.
  4. Eligible presbyopes will be those that wear full distance contact lenses in both eyes, then wear reading glasses over them.
  5. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of DW per day, at least 5 days per week, for a minimum of 1 month prior to the study) and willing to wear the study lenses on a similar basis.
  6. Subjects must be able and willing to wear the study lenses at least 6 hours a day, a minimum of 5 days per week.
  7. The subject's vertex-corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 (inclusive) in each eye.
  8. The subject's refractive cylinder must be ≤ -1.00 D in each eye.
  9. Have spherocylindrical best corrected visual acuity of 20/25+3 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other bodily diseases or infections, by self-report, which are known to interfere with contact lens wear and/or participation in the study.
  3. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear. Habitual medications taken by successful contact lens wearers are generally considered acceptable.
  4. Habitual toric, extended wear, or multifocal contact lens wear.
  5. Any current use of ocular medication.
  6. Any known hypersensitivity or allergic reaction to Optifree PureMoist.
  7. Any previous, or planned (during the course of the study) ocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  8. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  9. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  10. Any active or ongoing ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  11. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA slit-lamp scale.
  12. Binocular vision abnormality or strabismus.
  13. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that would contraindicate contact lens wear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - VRC-West, Foster City, California
  - Bartram Eye Clinic, Jacksonville, Florida
  - Pickens Family Eye Care, Pickens, South Carolina
  - Optometry Group, LLC, Memphis, Tennessee
  - William J. Bogus, OD, FAAO, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 92 subjects were enrolled into this study. Of those enrolled, 91 were dispensed a study lens and 1 subject failed to meet the eligibility criteria. Of the dispensed subjects 83 completed the study while 8 subjects were discontinued.
Groups:
- Test/Control/Control: Subjects that wore the Test lens during the first period, the Control lens during the second period and the Control lens again in the third period.
- Control/Test/Test: Subjects that wore the Control lens during the first period, the Test lens during the second period and the Test lens again in the third period.
Period: Period 1
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 46 | 45
Completed | 43 | 44
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 2 | 1
Period: Period 2
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 43 | 44
Completed | 40 | 43
Not Completed | 3 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 0 | 1
Period: Period 3
Arm/Group | Test/Control/Control | Control/Test/Test
Started | 40 | 43
Completed | 40 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Native Alaska | 0
  Asian | 11
  Black or African American | 3
  Native Hawaiian or Other Pacific Islander | 1
  White | 69
  Other | 7
Region of Enrollment [Number; unit: Participants]
  United States | 91

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Score
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. Observations from each study period are treated as independent (for the descriptive summary only). The average of all observations for each lens was reported.
Time Frame: 2- Week Follow-up Evaluation
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Test: Subjects that wore the Test lens during any of the three study periods.
- Control: Subjects that wore the Control lens during any of the three study periods.
Arm/Group | Test | Control
Number analyzed (Participants) | 78 | 78
Units on a scale | 61.49 (21.087) | 67.27 (22.865)
Statistical Analysis 1: Comparison: Test vs Control; It was calculated that 80 participants randomized in a 1:1 fashion between the two sequences would have at least 90% power to detect a 5 points difference in mean overall comfort at the 2-week follow-up. Sample size was determined using Stroup's Method (alpha=0.05); Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Linear Mixed Model; Kenward and Roger Method was used for the Degrees of Freedom; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-7.7 to -0.9], Standard Error of Mean 1.73 — Mean difference was calculated as Test - Control

2. Primary Outcome: Overall Vision Score
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. Observations from each study period are treated as independent (for the descriptive summary only). The average of all observations for each lens was reported.
Time Frame: 2- Week Follow-up Evaluation
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 78 | 78
Units on a scale | 61.79 (17.758) | 64.92 (17.444)
Statistical Analysis 1: Comparison: Test vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — A non-inferiority margin of -5 points was used. This margin is based on a 10% shift in the distribution of CLUE scores; Linear Mixed Model; Kenward and Roger Method was used for the Degrees of Freedom; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.7 to 1.0], Standard Error of Mean 1.43 — Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 6 weeks per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 0/91 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT03475875/Prot_SAP_000.pdf